CLINICAL TRIAL: NCT00921089
Title: The Association Among Vascular Calcification, Inflammation and Coronary Flow Velocity in Hemodialysis Patients
Brief Title: Vascular Calcification, Inflammation and Coronary Flow Velocity in Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Alaattin Yildiz, Istanbul Faculty of Medicine, Istanbul University
Other Study IDs: 1926
Record Dates: First submitted 2009-06-15; First posted 2009-06-16 (Estimated); Last update posted 2009-06-17 (Estimated); Status verified 2009-06

CONDITIONS: Renal Dialysis; Cardiovascular Diseases; Atherosclerosis; Inflammation
Keywords: Atherosclerosis; Cardiovascular disease; Hemodialysis; Inflammation; Vascular calcification
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis; Inflammation; Vascular Calcification

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hemodialysis group: End stage renal disease patients aged lower than 70 years, treated for more than 6 months with hemodialysis
- Control group: Normotensive healthy controls

SUMMARY:
The aim of this cross-sectional study is to determine the correlation of coronary artery calcification as measured by electron-beam computerized tomography and coronary flow reserve measured by trans-thoracic Doppler echocardiography in hemodialysis patients. The investigators also assessed the carotid artery parameters by measuring intima media thickness that can accurately describe the process of arterial wall changes due to atherosclerosis. Possible association of coronary flow reserve with inflammation and arterial calcification in hemodialysis patients was also evaluated.

DETAILED DESCRIPTION:
Cardiovascular mortality is a major cause of death in end-stage renal disease (ESRD). Therefore, the identification of coronary artery disease (CAD) in ESRD is an important task for nephrologists. Coronary angiography is the gold standard for detecting extent and severity of coronary atherosclerosis. It was necessary to determine whether coronary angiography, which is an invasive and contrast using procedure, should be performed in all high-risk individuals or whether noninvasive testing could reliably identify patients with critical coronary lesions. The coronary artery calcification (CAC) in uremic patients undergoing hemodialysis reflects the severity of atherosclerotic vascular disease and predicts the cardiovascular events. Recent studies of chronic kidney disease (CKD) patients have shown significant incidence and rapid progression rates of CAC. Coronary electron-beam computerized tomography (EBCT) could be used as screening test to identify cardiovascular disease (CVD) in CKD patients. In coronary artery disease, left ventricular diastolic dysfunction was found to be correlated with reduced coronary flow reserve (CFR) in patients with hypertension and left ventricular hypertrophy. This shows that in patients with vascular calcification, CFR measurement by trans-thoracic Doppler echocardiography (TTDE) as a non-invasive and an easy test has a usage advantage during risk stratification. CFR represents the capacity of the coronary circulation to dilate following an increase in myocardial metabolic demands. By using this method, impairment of CFR can be assessed before development of angiographically detectable stenosis in epicardial coronary arteries and we are able to investigate early coronary microvasculature pathology. The aim of this cross-sectional study, is to determine the correlation of CAC as measured by EBCT and CFR measured by TTDE. We also assessed the carotid artery parameters by measuring intima media thickness that can accurately describe the process of arterial wall changes due to atherosclerosis. Possible association of CFR with inflammation and arterial calcification was also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 years of age or older and able to give informed consent
* End stage renal disease patients treated for more than 6 months with hemodialysis

Exclusion Criteria:

* Valvular heart disease
* Prior myocardial infarction
* Any prior coronary intervention
* Dilated or hypertrophic cardiomyopathy
* Congestive heart failure
* Cardiac arrhythmia
* Active infection or non-infectious overt inflammation
* Patients whose LAD could not visualized adequately

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: End stage renal disease patients and normotensive healthy controls were studied for the assessment of coronary artery calcification score by electron-beam computerized tomography and coronary flow reserve trans-thoracic Doppler harmonic echocardiographyby.
Sampling Method: Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2008-04; Primary Completion 2008-07 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Comparison of coronary artery calcium scores measured by electron-beam computerized tomography and coronary flow reserve. | 3 months

SECONDARY OUTCOMES:
Relationship between coronary artery calcium scores, coronary flow reserve and inflammatory parameters (IL-6,TNF-alpha, hs-CRP). | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Alaattin Yildiz, MD, Study Director — Division of Nephrology, Istanbul Faculty of Medicine, Istanbul University; Yasar Caliskan, MD, Principal Investigator — Division of Nephrology, Istanbul Faculty of Medicine, Istanbul University
Locations (1):
- Division of Nephrology, Department of Internal Medicine, Istanbul Faculty of Medicine, Istanbul University, Istanbul, Turkey (Türkiye)